CLINICAL TRIAL: NCT05683301
Title: Treatment Optimisation for Blood Pressure With Single-Pill Combinations in India
Acronym: TOPSPIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Chronic Disease Control, India (Other)
Collaborators: All India Institute of Medical Sciences (Other); Imperial College London (Other)
Responsible Party: Principal Investigator, Dr. Dorairaj Prabhakaran, Executive Director, Centre for Chronic Disease Control, India
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CCDC-2022-001
Record Dates: First submitted 2022-12-10; First posted 2023-01-13 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Primary Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — amlodipine, perindopril drug combination; indapamide, perindopril drug combination; Amlodipine; Indapamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): (Arm 1 compare to Arm 2 compare to Arm 3) - Treatment Period 1 (Enrollment - 2 months) - Single Pill Combination of Amlodipine 5 mg and Perindopril 4 mg once daily, orally Treatment Period 2 (2 months - 6 months) - Single Pill Combination of Amlodipine 10 mg and Perindopril 8 mg once daily, orally
  Interventions: Drug: Amlodipine + Perindopril
- Arm 2 (Experimental): (Arm 1 compare to Arm 2 compare to Arm 3) - Treatment Period 1 (Enrollment - 2 months) - Single Pill Combination of Perindopril 4 mg and Indapamide 1.25 mg once daily, orally Treatment Period 2 (2 months - 6 months) - Single Pill Combination of Perindopril 8 mg and Indapamide 2.5 mg once daily, orally
  Interventions: Drug: Perindopril + Indapamide
- Arm 3 (Experimental): (Arm 1 compare to Arm 2 compare to Arm 3) - Treatment Period 1 (Enrollment - 2 months) - Single Pill Combination of Amlodipine 5 mg and Indapamide 1.5 mg sustained release once daily, orally Treatment Period 2 (2 months - 6 months) - Single Pill Combination of Amlodipine 10 mg and Indapamide 1.5 mg sustained release once daily, orally
  Interventions: Drug: Amlodipine + Indapamide

INTERVENTIONS:
Drug: Amlodipine + Perindopril — Single pill combination of dual antihypertensive agent
  Arms: Arm 1
Drug: Perindopril + Indapamide — Single pill combination of dual antihypertensive agent
  Arms: Arm 2
Drug: Amlodipine + Indapamide — Single pill combination of dual antihypertensive agent
  Arms: Arm 3

SUMMARY:
Hypertension is a leading cause of morbidity and mortality globally. Although multiple drugs are frequently used to treat it, in the South Asian context, evidence is lacking on best drug combinations. This trial aims to compare efficacy of three single-pill combinations of two anti-hypertensive agents on 24-hour ambulatory systolic blood pressure among 1968 individuals with hypertension. The trial is a single-blind randomized controlled trial spread across 37 hospitals in India.

Single Pill combinations (SPCs): 1) Amlodipine + Perindopril, 2) Perindopril + Indapamide, 3) Amlodipine + Indapamide

DETAILED DESCRIPTION:
This is a multi-centre, individual randomized single-blind, parallel group, three-armed superiority trial to compare the efficacy of three different single-pill combinations of antihypertensive therapies (Amlodipine/Perindopril, Perindopril/Indapamide, and Amlodipine/Indapamide)on 24-hour ambulatory BP levels in Indians.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30-79 years AND
2. Sitting clinic values* of SBP ≥140 mmHg and <160 mmHg on one antihypertensive agent OR
3. Sitting clinic values* of SBP ≥150 mmHg and <180 mmHg on no antihypertensive treatment * Mean of the last 2 of 3 readings.

Exclusion Criteria:

1. Congestive heart failure (clinically defined).
2. Patients with a history of intolerance to any of the study medications for example angioedema or dry cough with Angiotensin-converting enzyme inhibitors.
3. Serum creatinine levels greater than 132.6µmol/l (1.5mg/dl)
4. 4. History of coronary heart disease (i.e., chronic stable angina, myocardial infarction or acute coronary syndrome).
5. History of a stroke or other cerebrovascular accident (i.e. transient ischaemic attack or reversible ischaemic neurological deficit).
6. Severe hepatic impairment
7. Treatment with agents causing torsades de pointes
8. Lactation
9. Contraindications to any of the investigational medicinal products as per the summaries product characteristics of drugs studied
10. Known or suspected secondary hypertension.
11. Any other concomitant illness, physical or mental impairment that could interfere with the effective conduct of the study.
12. Pregnancy or those of child-bearing age who are not taking reliable contraception.
13. History of Gout.
14. Serum potassium < 3.5mmol/L at screening.

    -

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1981 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-09-22 (Actual)

PRIMARY OUTCOMES:
24-hour ambulatory systolic Blood Pressure | Change in between baseline and 6 month Ambulatory Systolic Blood Pressure
  To determine which of three single pill combinations of two anti-hypertensive agents is most effective in reducing 24-hour ambulatory systolic BP (ASBP) in Indian patients with hypertension.

SECONDARY OUTCOMES:
24-hour ambulatory diastolic blood pressure | Change in between baseline and 6 month Ambulatory Diastolic Blood Pressure
  To determine which of three single pill combinations of two antihypertensive agents is most effective in reducing 24-hour ambulatory diastolic blood pressure at 6 months adjusted for baseline ADBP
Clinic Blood Pressure | Comparison of Clinic blood pressure measured at baseline 2 month , 4 month and 6 month
  To determine which of three single pill combinations of two antihypertensive agents is most effective in reducing Clinic SBP and diastolic blood pressure (DBP) at two, four and six months adjusted for baseline values
Daytime and nighttime Blood Pressure | Change in between baseline and 6 month ASBP and ADBP
  To determine which of three single pill combinations of two antihypertensive agents is most effective in reducing Daytime and nighttime blood pressure (BP) a t six months adjusted for baseline values
BP variability measured by ABPM and within-visit clinic BPs | Fluctuations in Ambulatory blood pressures as measured at baseline and 6 month and fluctuation in Clinic BP as measured at baseline, 2 month, 4 month and 6 month
  To determine which of three single pill combinations of two antihypertensive agents is most effective in reducing 3.2.4. BP variability measured by ASBP and within-visit clinic BP
Proportion of patients who achieve BP control | BP control measured in Clinic BP as measured at baseline, 2 month, 4 month and 6 month and ABP measured at baseline and 6 month
  To determine which of the three single pill combinations of two antihypertensive agents is most effective in increasing the proportion of patients who achieve BP control defined as BP: <140/90 mmHg and <130/80mmHg at any of their clinic visits and maintained at the 6-month clinic visit.
Proportion of patients classified as "responders" | Clinic BP as measured at baseline, 2 month, 4 month and 6 month
  Proportion of patients classified as "responders" defined as those who had a reduction of SBP ≥20mmHg and DBP ≥10 mmHg at any of their clinic visits and maintained at the 6-month clinic visit.
Micro- and macro-albuminuria | Change in serum albumin measured at baseline and 6 month
  To determine the effect of three single pill combinations of two antihypertensive agents on Micro- and macro-albuminuria.
Fasting blood glucose | Change in fasting blood glucose measured at baseline and 6 month
  To determine the effect of three single pill combinations of two antihypertensive agents on Fasting blood glucose.
Fasting lipid profile | Change in serum lipid profile measured at baseline and 6 month
  To determine the effect of three single pill combinations of two antihypertensive agents on fasting lipid profile.
Serum sodium | Change in serum sodium measured at baseline and 6 month
  To determine the effect of three single pill combinations of two antihypertensive agents on serum sodium
Serum potassium | Change in serum potassium measured at baseline and 6 month
  To determine the effect of three single pill combinations of two antihypertensive agents on serum potassium
Serum urea | Change in serum urea measured at baseline and 6 month
  To determine the effect of three single pill combinations of two antihypertensive agents on serum urea
Serum creatinine | Change in serum creatinine measured at baseline and 6 month
  To determine the effect of three single pill combinations of two antihypertensive agents on serum creatinine
eGFR | Change in eGFR measured at baseline and 6 month
  To determine the effect of three single pill combinations of two antihypertensive agents on eGFR
Adverse events causing trial withdrawal | adverse events causing withdrawal at 2 month, 4 month and 6 month
  To determine the effect of three single pill combinations of two antihypertensive agents on adverse events causing trial withdrawal
renin and aldosterone | Change in plasme renin and/or aldosterone measured at baseline and 6 month
  To determine whether baseline plasma renin and/or aldosterone predicts any differential BP effects of the three single-pill combinations under investigation.

CONTACTS AND LOCATIONS:
Overall Officials: Dorairaj Prabhakaran, DM Cardiology, Principal Investigator — Centre for Chronic Disease Control, New Delhi
Locations (35):
- India (35):
  - Lalitha Super Specialities Hospital, Guntur, Andhra Pradesh
  - Apollo Hospitals, Visakhapatnam, Andhra Pradesh
  - Assam Medical College, Dibrugarh, Assam
  - Apollo-Excelcare Hospital, Guwahati, Assam
  - Rudraksha Hospital, Ahmedabad, Gujarat
  - Apollo Hospitals, Ahmedabad, Gujarat
  - Aman Hospital & Research Center, Vadodara, Gujarat
  - Lifecare Hospital & Research Centre, Bangalore, Karnataka
  - SDM College of Medical Sciences & Hospital, Dharwad, Karnataka
  - Indiana Hospital & Heart Institute, Mangalore, Karnataka
  - JSS Hospital, Mysore, Karnataka
  - BLDE, Shri B. M. Patil Medical College, Hospital & Research Centre, Vijayapura, Karnataka
  - Lisie Hospital, Ernākulam, Kerala
  - Lakshmi Hospital, Palakkad, Kerala
  - BKL Walawalkar Rural Medical College and Hospital, Devran, Maharashtra
  - Bhatia Hospital, Mumbai, Maharashtra
  - Sengupta Hospital & Research Institute, Nagpur, Maharashtra
  - Shalinitai Meghe Hospital and Research Center, Nagpur, Maharashtra
  - Nazareth Hospital, Shillong, Meghālaya
  - North Eastern Indira Gandhi Regional Institute of Medical Sciences, Shillong, Meghālaya
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Indraprastha Apollo Hospitals, New Delhi, National Capital Territory of Delhi
  - Apollo Hospitals, Bhubaneshwar, Odisha
  - All India Institute of Medical Sciences, Bathinda, Punjab
  - Dayanand Medical College and Hospital, Ludhiana, Punjab
  - Sadbhavna Medical and Heart Institute, Patiāla, Punjab
  - SP Medical College, Bikaner, Rajasthan
  - All India Institute of Medical Sciences, Jodhpur, Rajasthan
  - Madras Medical College, Chennai, Tamil Nadu
  - Sri Ramchandra Institute of Higher Education and Research, Chennai, Tamil Nadu
  - Apollo Hospital, Madurai, Tamil Nadu
  - Osmania General Hospital, Hyderabad, Telangana
  - Apollo DRDO Hospitals, Hyderabad, Telangana
  - Apollo Institute of Medical Sciences, Hyderabad, Telangana
  - Mediciti Institute of Medical Sciences, Hyderabad, Telangana

IPD SHARING:
Plan to Share IPD: Yes
De-identified data collected for the study will be shared with bonafide researchers with a valid research question. Request may be addressed to Prof. Prabhakaran - dprabhakaran@ccdcindia.org
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 01-09-2025 till 30-09-2030
Access Criteria: Only bonafide researchers with a valid research question shall be provided data. Interested researchers shall write to Prof. Prabhakaran (dprabhakaran@ccdcindia.org) with a concept note and necessary approvals as applicable.

REFERENCES:
- [Derived] Prabhakaran D, Roy A, Chandrasekaran AM, Kondal D, Mukherjee S, Kiru G, Singh K, Salwa H, Sobitharaj EC, Lobo AS, Mahajan G, Mohan B, Khanna A, Malviya A, Patil SG, Abichandani VK, Singh B, Gupta BK, Yellapantula B, Dandge S, Sengupta S, Kumar S, Bardoloi N, Senguttuvan NB, Sahay RK, Patil S, Deora S, Prahalad R, Sarvepalli VP, Gnanaraj JP, Khanna M, Mishra A, Aithal K, Chavda V, Cornelius VR; TOPSPIN Clinical Consortia; Poulter NR. Comparison of dual therapies for hypertension treatment in India: a randomized clinical trial. Nat Med. 2025 Sep;31(9):3169-3175. doi: 10.1038/s41591-025-03854-w. Epub 2025 Jul 25. PMID 40715816